CLINICAL TRIAL: NCT01984411
Title: Comparison of Vascular ACcess for Radial and Femoral Completion of Diagnostic Cardiac Catheterization Performed at the Clinic Patients Northern General de Barranquilla in 2013. Controlled Clinical Trial of Non-inferiority
Brief Title: Comparison of Vascular Access for Radial and Femoral Completion of Diagnostic Cardiac Catheterization
Acronym: COMPACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Cardiológico del Caribe, Columbia (Other)
Responsible Party: Principal Investigator, Celin Malkun, Cardiologist Interventional, Centro Cardiológico del Caribe, Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCCColumbia
Record Dates: First submitted 2013-10-25; First posted 2013-11-14 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Ischemic Heart Diseases
MeSH Terms: conditions — Myocardial Ischemia | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radial Technical (Experimental): Radial technical is the procedure for catheterization
  Interventions: Procedure: Radial Technical; Drug: Omnipaque
- Femoral Technical (Active Comparator): Vascular Access for cardiac catheterization
  Interventions: Procedure: Femoral Technical; Drug: Omnipaque

INTERVENTIONS:
Procedure: Radial Technical — Vascular Access for cardiac catheterization
  Arms: Radial Technical
Procedure: Femoral Technical — Vascular Access for cardiac catheterization
  Arms: Femoral Technical
Drug: Omnipaque
  Other Names: Iohexol

SUMMARY:
Cardiac catheterization is the most important test for the evaluation of cardiac patients. Since the beginning of the cardiac catheterization procedure, we have used the femoral artery puncture as a gateway for those procedures. Recently it is used more often the path for the radial. Using this approach has gained many followers worldwide and has been used almost routinely in our country but has not gained popularity because many interventional cardiologists argue that the transradial procedure is much more time-consuming and difficult.

Research question: Are there differences in the total procedure time path between radial and femoral vascular to perform cardiac catheterizations?.

This research focuses on the search for information to determine whether there are significant differences when the variables under study. This research is justified by the need to evaluate the two techniques in use and the lack of studies evaluating and comparing the radial arterial access in comparison with femoral access route which is widely used in all services hemodynamics national and international. The lack of research on the subject has made the use of the transradial procedure routinely not being done, because they have the idea that it is much more time-consuming and technically more difficult than the procedure performed by the femoral approach, hence Hemodynamics specialists, not everyone wants to start implementing the systematic use of the radial approach for cardiac catheterization studies.The main objective of this project is to determine the non-inferiority in terms of total procedure time path between radial and femoral vascular to perform cardiac catheterizations. Secondary objectives: the difference in time of puncture, duration of the procedure and recovery. Incidence of vascular complications and techniques between radial and femoral, presence of complications at 8 days of follow-up. Our aims to check through the results, if the difference in each of the variables favoring either of the two techniques and to determine the non-inferiority of one technique over the other in terms of ease and effectiveness of both procedures. The type of study is a controlled clinical trial open, randomized, non-inferiority. The study population will consist of patients who have been told the diagnostic cardiac catheterization, they are sent to the General Clinic Northern institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients requiring a performing diagnostic cardiac catheterization procedure, scheduled electively or urgently,
* Patients mentally healthy
* Patients with test Allen (palmar arch patency) normal
* Patients who signing the informed consent.

Exclusion Criteria:

* Patients with a history of allergic reaction to the dye.
* Patients with peripheral vascular disease.
* Anticoagulated patients with coumarinic or other oral anticoagulants.
* Patients with arteriovenous fistula for hemodialysis.
* Patients with a history of coronary artery bypass surgery.
* Patients with amputations or upper limb deformities.
* Patients with limited movement in the upper limbs or burns contractures.
* Patients requiring catheterization while the right heart do.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Minutes Total Procedure Time | Assess the total duration of the procedure in minutes. Up to 15 min
  The primary outcome measure in this trial, is the time in minutes spent on the realization of the entire cardiac catheterization procedure

SECONDARY OUTCOMES:
Minute of Fluoroscopic time | Assess the total duration of the procedure in minutes. Up to 5 min
  This secindary outcome is the time in minutes spent during fluoroscopy

OTHER OUTCOMES:
Complications | 8 days
  Vascular and Clinical complications

CONTACTS AND LOCATIONS:
Overall Officials: Celin Malkun, MD, MSc, Principal Investigator — Centro Cardiológico del Caribe, Columbia; Jorge Luis Acosta, MD, MSc, Study Director — Universidad del Norte, Barranquilla, Colombia
Locations (1):
- Clinica General del Norte, Barranquilla, Atlco, Colombia